CLINICAL TRIAL: NCT03855202
Title: The Treatment of Bronchopulmonary Dysplasia by Instillation PS and Mononuclaer Cells in Preterms
Acronym: BPD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: yangjie (Other)
Responsible Party: Sponsor-Investigator, yangjie, Director of Dept of Neonatology, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Guangdong W C H
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Neonates Premature; Ventilator Support
Keywords: PS; cord blood mononuclaer Cells; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- infusion froup 1 (Experimental): autologuous umbilical cord blood mononuclear cells 48 hours after birth ,dose is 25 million cells/kg
  Interventions: Biological: CBMNC
- infusion group 2 (Experimental): autologuous umbilical cord blood mononuclear cells 48 hours after birth ,dose is 25 million cells/kg ,PS,dose is 70mg/kg
  Interventions: Biological: PS+CBMNC
- infusion group 3 (Experimental): PS,dose is 70mg/kg
  Interventions: Biological: PS
- Placebol (Placebo Comparator): 0.9% sodium chloride installation after 24 hours
  Interventions: Other: Placeo

INTERVENTIONS:
Biological: CBMNC — autologuous umbilical cord blood mononuclear cells 48 hours after birth ,dose is 25 million cells/kg
  Arms: infusion froup 1
Biological: PS+CBMNC — autologuous umbilical cord blood mononuclear cells 48 hours after birth ,dose is 25 million cells/kg ,PS,dose is 70mg/kg
  Arms: infusion group 2
Biological: PS — PS,dose is 70mg/kg
  Arms: infusion group 3
Other: Placeo — 0.9% sodium chloride installation after 24 hours
  Arms: Placebol

SUMMARY:
Bronchopulmonary dysplasia mainly occurs in premature infants, which is the main cause of premature infant death.If children with BPD can survive, they are also prone to complications of long-term respiratory diseases such as asthma,that affect the quality of life of BPD children. However, there is no effective treatment method for BPD. So,the investigator would like to investigate the effect of Intratracheal PS and mononuclaer cells in pretems

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial that constitues one time points cohor and three group,each group with 80 participants,which receive intratracheal PS and mononuclaer cells,receive intratracheal PS,receive intratracheal mononuclaer cells.

1. Eligibility Criteria:Preterm(gestational age more than 28weeks and less than 37weeks)
2. Exlusion criteria: Preterm infants with major congenital malformations,chromosomal anomalies,inborn errors of metabolism and clinical or laboratory evidence of a congenital infection
3. Demographic Data and Baseline characteristics of the study groups were collected:

Gestational age(weeks) birth weight(g) gender Cesarean section delivery antenatal steroids prolonged rupture of membrane Multiple pregnancies APGAR score at 5 minutes Thrombocytopenia before intervention CRP befor intervention(mg/l) TNF-αbefore intervention（pg/ml） 4.Autologous cord blood mononuclear cells doses is 25million cells/kg 5.the following are monitored at 3、7、14、21 days after birth: mortality, incidence of bronchopulmonary dysplasia 5.Long-term follow up:in 1m，3m，6m,1y:neurodevelopment,asthma，anemia and physic growth

ELIGIBILITY:
Inclusion Criteria:

twenty-eight weeks to thirty-seven weeks

Exclusion Criteria:

Pretem infants with major congenital malformations,chromosomal anomalies,inborn errors of metabolism and clinical or laboratory evidence of a congenital infection

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2019-02-24 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
number of patients who died | up to 21 days after birth
  mority rate

SECONDARY OUTCOMES:
number of patients with neurodevelopmental disorder assessed by Bayley Score | up to 1 month, 3 month, 6 months and 1 year
  Long term follow up:in 1 month, 3months,6 months,and 1 years:

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Guangdong Women and Children Hospital

IPD SHARING:
Plan to Share IPD: No